CLINICAL TRIAL: NCT03541265
Title: Efficacy of Regional Adductor Canal Block Using Extended Release Liposomal Bupivacaine in Total Knee Arthroplasty: A Randomized Prospective Study
Brief Title: Liposomal Bupivacaine in Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bronx-Lebanon Hospital Center Health Care System (Other)
Responsible Party: Principal Investigator, Morteza Meftah, Chief, Adult Recosntruction Orthopaedic Surgery, Bronx-Lebanon Hospital Center Health Care System
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 04141603
Record Dates: First submitted 2018-04-25; First posted 2018-05-30 (Actual); Last update posted 2018-05-30 (Actual); Status verified 2018-05

CONDITIONS: Knee Osteoarthritis; Anesthesia, Local
Keywords: liposomal bupivacaine; total knee arthroplasty
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: This is a a randomized prospective study. Patients were assigned into two cohorts on the day of surgery using a randomization software by an independent observer. Randomization was based on age, gender, BMI and type of surgery. The investigators hypothesized that there would be no difference in the pain scores or morphine consumption. Sample size analysis for a randomized prospective trial was performed to achieve an 80% power to detect 20% difference in pain scores (2-point score difference on VAS 0-10 was deemed clinically relevant). A sealed envelope was given to the anesthesiologist and the surgeon on the day of surgery, stating the group that the patient was assigned to participate. All descriptive statistics (Mean, SD) and analysis were performed with SPSS version 21 (IBM) at a 0.05 level of significance.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Adductor block protocol (Experimental): An ultrasound-guided injection of Subsartorial saphenous nerve using Exparel 266 mg (20 cc vial) via a 21-gauge 4-inch Stimuplex A needle (B. Braun Medical Inc., Melsungen, Germany) was performed at mid-thigh level with a high-frequency linear ultrasound transducer. All regional anesthesia was performed by a trained anesthesiologist. Ultrasound pictures (pre-injection and post-injection) was obtained to verify proper local anesthetic placement.
  Interventions: Drug: Exparel; Procedure: Adductor block protocol
- peri-articular injection (Active Comparator): Peri-articular injection included combination of Exparel 266 mg (20 ml vial) with 20 ml of 0.5% bupivacaine, and normal saline to a total volume of 120 ml. The injection was meticulously administered prior and after cementation in the posterior capsule, posteromedial structures, the periarticular synovium, extensor apparatus, pes anserinus, anteromedial capsule, periosteum, iliotibial band, and subcutaneous plane. Injections were performed using 20-mL syringes with 22-gauge needle, minimal leakage. Visible tissue expansion was achieved.
  Interventions: Drug: Exparel; Procedure: peri-articular injection protocol

INTERVENTIONS:
Drug: Exparel — long-acting Bupivacaine extended release liposome compound
  Other Names: Liposomal Bupivacaine
Procedure: Adductor block protocol — Adductor block using Exparel
  Arms: Adductor block protocol
Procedure: peri-articular injection protocol — peri-articular injection using Exparel
  Arms: peri-articular injection

SUMMARY:
Pain management after total knee arthroplasty is essential for optimized clinical outcomes and higher satisfaction. Exparel (Pacira Pharmaceuticals, Parsippany, New Jersey, USA) is a long-acting Bupivacaine extended release liposome compound that is injected peri-articularly or as regional block. The purpose of this study was to compare the analgesic efficacy of single administration of Exparel for local peri-articular infiltration versus adductor canal regional block.

DETAILED DESCRIPTION:
Multimodal pain approach is now an accepted standard of care to improve pain, enable earlier mobilization and faster recovery, decreased length of stay, and reduce opioid consumption and related side effects. The multimodal approach includes peri-operative oral and IV analgesics, local periarticular injections (PAI), and/or regional blocks such as femoral nerve blocks nerve or subsartorial saphenous nerve (adductor canal) blocks. Extended release bupivacaine (Exparel - Pacira Pharmaceuticals, Parsippany, NJ, USA) in liposomal form was developed for longer lasting post-operative analgesia. There are limited studies analyzing its efficacy of single injection liposomal bupivacaine in adductor canal block in total knee arthroplasty. The investigators hypothesized that a single adductor canal regional block injection would provide similar pain relief as peri-articular infiltration of Exparel.

ELIGIBILITY:
Inclusion Criteria:

* primary knee osteoarthritis undergoing unilateral knee replacement

Exclusion Criteria:

* hypersensitivity and/or allergies to local anesthetics or previous knee surgery

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2018-03-01 (Actual)

PRIMARY OUTCOMES:
Difference in mean pain scores in the first 3 days after surgery | 3 days
  Pain was recorded during the first 3 post-operative days after surgery on scale 0 to 10 (visual analog scale). Zero represents 'no pain', as the best outcome and 10 represents as 'the worst pain experienced' as the worst outcome.The difference between the mean pain score in the two groups is assessed.

SECONDARY OUTCOMES:
Difference in mean opioid consumption in the first 3 days after surgery | 3 days
  All opioids were converted to Morphine equivalent consumption (MEC) during the first 3 days. The difference in the mean MEC in the two groups is assessed.